CLINICAL TRIAL: NCT01367730
Title: Non-Invasive Assessment of Bone Micro-architecture and Strength Changes in Men With Osteopenia and Osteoporosis
Brief Title: Assessment of Bone Micro-Architecture Using HR-pQCT
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Majumdar #39637
Record Dates: First submitted 2011-06-02; First posted 2011-06-07 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Osteoporosis
Keywords: osteopenia and osteoporosis
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- osteoporosis and osteopenia: Subjects will be stratified based on DXA BMD T-scores.

SUMMARY:
In the context of male osteoporosis, we hypothesize that regional changes in trabecular bone, as well as changes in cortical porosity will play a major role, and thus also affect bone strength. In developing therapeutics the response of individual compartments, regional variations post-therapy will have considerable impact on selecting the therapies as well as monitoring response to therapy. This study, a precursor to other therapeutic trials, will lay the ground-work for the future.

DETAILED DESCRIPTION:
We will recruit 80 subjects who will be stratified into groups based on their T-scores. All subjects will be imaged at Baseline and 12 months. Measures of bone micro-architecture in the tibia and radius using peripheral computed tomography, bone strength measures through finite element analysis will be obtained at all time points. DXA measures at the spine, femur and forearm will be obtained as reference measures. In addition whole body DXA scans will be performed for assessment of body composition.

ELIGIBILITY:
Inclusion Criteria:

1. Men 50-85 years old
2. Patients must be willing to undergo a DXA scan.
3. Patients should be willing to undergo HRpQCT scan of the radius and tibia.

Exclusion Criteria:

1. Inability to tolerate CT scans
2. Use of medications known to impact bone and mineral metabolism:

   * use of a bisphosphonate or teriparatide in the last year or for >12 months ever;
   * current calcitonin;
   * prednisone >5 mg daily or the equivalent glucocorticoid for >10 days in the last 3 months;
   * current testosterone therapy;
   * current thiazolidinedione (TZD);
   * current androgen deprivation therapy;
   * current use of an antiepileptic agent that alters hepatic vitamin D clearance;
   * use of thyroid hormone replacement with current thyroid stimulating hormone <0.1 mIU/L
3. Disease known to affect bone (e.g., primary hyperparathyroidism, Pagets disease, clinically significant liver disease)
4. Illicit drug use or alcohol use >3 drinks/day
5. Serum calcium >10.2 mg/dL or calculated creatinine clearance <30 mL/min
6. Weight >350 pounds (the maximum weight limit of the DXA)
7. Hardware in the lumbar spine
8. History of bilateral hip replacement, or bilateral wrist or ankle fracture

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community UCSF VA Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Measure cross-sectional and longitudinal differences in bone micro-architecture and strength changes in men with BMD T-scores ≤-2.0 and those with T-scores >-1.0. | 12 months
  Trabecular bone micro-architecture as measured by trabecular number, trabecular BMD, and trabecular bone volume fraction (BV/TV). Cortical bone micro-architecture will be assessed by measuring cortical density & thickness and porosity.

SECONDARY OUTCOMES:
Change in Compressive biomechanical bone properties from Baseline to 12 months | 12 months
  Calculate the change in compressive biomechanical properties using µ-finite element analysis
Association between BMD, bone micro-architecture, compressive biomechanical properties and body composition at all timepoints | Baseline and 12 months
  Association between BMD, bone micro-architecture, compressive biomechanical properties and body composition at all timepoints using DXA, HR-pQCT, microfinite element analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Majumdar, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Imaging Center, San Francisco, California, United States